CLINICAL TRIAL: NCT05712460
Title: A PHASE 1, RANDOMIZED, SPONSOR OPEN, TWO-PART CROSSOVER STUDY TO ASSESS SAFETY, TOLERABILITY, PHARMACOKINETICS AND FOOD EFFECT OF MULTIPLE DOSES IN PART 1 AND PALATABILITY OF A SINGLE DOSE OF SISUNATOVIR IN PART 2, IN HEALTHY ADULT PARTICIPANTS
Brief Title: A Study to Assess the Safety, Effects and Palatability of Sisunatovir in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: C5241006; 2022-003426-53 (EudraCT Number)
Record Dates: First submitted 2023-01-25; First posted 2023-02-03 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Respiratory Syncytial Viruses
Keywords: RSV; respiratory syncytial virus
MeSH Terms: interventions — sisunatovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group A: Higher dose sisunatovir (Experimental): higher dose of sisunatovir dosed every 12 hours
  Interventions: Drug: sisunatovir
- Group B: Lower dose sisunatovir (Experimental): Lower dose of sisunatovir dosed every 12 hours
  Interventions: Drug: sisunatovir
- Group C: Placebo (Placebo Comparator): Placebo for sisunatovir dosed every 12 hours
  Interventions: Drug: Placebo
- Group D: Higher dose of sisunatovir (Experimental): Higher dose of sisunatovir dosed every 12 hours under fasted conditions
  Interventions: Drug: sisunatovir
- Group E: sisunatovir palatability (Experimental): Sisunatovir in 4 vehicles (water, saline, apple juice, infant formula) to assess the palatability of sisunatovir in each vehicle. sisunatovir will not be swallowed, participants will swirl and spit to assess various aspects of the taste.
  Interventions: Drug: sisunatovir

INTERVENTIONS:
Drug: sisunatovir — Sisunatovir is an orally administered RSV F-protein inhibitor being developed to target viral-host cell fusion for the treatment of adult and pediatric patients with RSV
  Arms: Group A: Higher dose sisunatovir; Group B: Lower dose sisunatovir; Group D: Higher dose of sisunatovir; Group E: sisunatovir palatability
Drug: Placebo — Placebo for sisunatovir
  Arms: Group C: Placebo

SUMMARY:
This study is seeking healthy participants who are:

1. Aged 18 to 65 years of age. All fertile participants must agree to use a highly effective method of contraception.
2. Male and female participants who are overtly healthy as determined by medical evaluation. This includes medical history, physical examination, blood pressure, pulse rate, standard 12-lead ECG (electrocardiogram), and laboratory tests.
3. BMI (body mass index) of 17.5 to 35 kg/m2; and a total body weight >50 kg (110 lb).

This study will consist of up to 2 cohorts (groups of participants).:

Cohort 1 is a randomized, 2-part, crossover cohort. Part 1 has 3 periods. Periods 1 and 2 are to evaluate the safety and effects of sisunatovir. Participants will take sisunatovir tablets or placebo by mouth once every 12 hours. A placebo looks like the study medicine but does not contain any active medicine in it.

Period 3 is an open label period to evaluate the food effect of the planned higher dose of sisunatovir. Participants will take the planned higher dose sisunatovir tablets every 12 hours. In Part 2, participants will take sisunatovir prepared in 4 different vehicles (water, infant formula, apple juice, and saline) to assess how palatable each form is. Participants will complete a questionnaire after tasting each form of sisunatovir. The palatability questionnaire will be completed for each vehicle, the questionnaire asks participants to assess each vehicle at 4 different time increments after tasting. At least 60 minutes will pass between tasting each vehicle. Period 4 may start after the last PK draw of Period 3.

A minimum 7-day washout period will occur between the last dose of Periods 1 and 2 and the first dose of Periods 2 and 3. We will assess the safety of participants following each study period and doses and adjust the doses for subsequent study periods as needed.

Cohort 2 is an optional cohort; the design of Cohort 2 is the same as Part 1 of Cohort 1. Dose levels studied in Cohort 2 will be determined after the completion of Cohort 1.

Participants will take part in this study for approximately 2 months, excluding the screening period. During this time there are 3 separate 7-day in-patient stays at the study clinic and a follow-up phone call that takes place 28-35 days after the last dose of study medicine.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 18 to 65 years of age, inclusive, at the time of signing of the informed consent document (ICD).

   • All fertile participants must agree to use a highly effective method of contraception.
2. Male and female participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, including blood pressure, pulse rate, standard 12-lead electrocardiogram (ECG), and laboratory tests.
3. Body mass index (BMI) of 17.5 to 35 kg/m2; and a total body weight >50 kg (110 lb).

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality, or other conditions or situations related to Coronavirus Disease 2019 (COVID-19) pandemic that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
3. Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention with the exception of moderate/strong CYP3A inducers or time dependent inhibitors which are prohibited within 14 days plus 5 half lives prior to the first dose of study intervention.
4. A positive urine drug test, confirmed by a repeat test, if deemed necessary.
5. Screening supine blood pressure (BP) ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest. If BP is ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
6. Standard 12 lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results.
7. Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary:

   * glomerular filtration rate (GFR) <60 mL/min/1.73m2 based on the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation;
   * Aspartate Aminotransferase (AST) or Alanine Transaminase (ALT) level ≥1.5 x upper limit of normal (ULN);
   * Gamma-glutamyl transferase (Gamma-GT)> ULN;
   * Alkaline phosphatase > ULN;
   * Total bilirubin level ≥1.5 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ ULN.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5241006

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was planned to be conducted in 2 cohorts: Cohort 1 and optional Cohort 2. Cohort 1 had 2 parts, Part 1 had 3 periods (Period 1, 2, 3) and Part 2 had 4 periods (Period 4, 5, 6, 7). The optional cohort 2 was not conducted based on the findings for Cohort 1.
Pre-assignment Details: A total of 12 participants were enrolled at 1 site in Brussels.
Groups:
- Treatment Sequence: ABDEFGH: Sisunatovir 400 mg, Fed (treatment A) was administered once every 12 hours (Q12h) for 4 days in Period 1, followed by sisunatovir 200 mg plus matching placebo, Fed (treatment B) Q12h for 4 days in Period 2 followed by sisunatovir 200 mg, Fasted (treatment D) administered Q12h for 4 days in Period 3. There was a washout period of minimum 7 days between each subsequent period. Participants tasted sisunatovir 50 mg capsule content in water (treatment E) followed by sisunatovir 50 mg in Formula (treatment F) sisunatovir 50 mg in apple juice (treatment G) and sisunatovir 50 mg in saline (treatment H) on Day 1 of treatment period 4 to 7. There was a washout of at least 60 minutes between tasting each vehicle.
- Treatment Sequence: ABDFGHE: Sisunatovir 400 mg, Fed (treatment A) was administered Q12h for 4 days in Period 1, followed by sisunatovir 200 mg plus matching placebo, Fed (treatment B) Q12h for 4 days in Period 2 followed by sisunatovir 200 mg, Fasted (treatment D) administered Q12h for 4 days in Period 3. There was a washout period of minimum 7 days between each subsequent period. Participants tasted sisunatovir 50 mg in Formula (treatment F) followed by sisunatovir 50 mg in apple juice (treatment G) and sisunatovir 50 mg in saline (treatment H), sisunatovir 50 mg capsule content in water (treatment E) on Day 1 of treatment period 4 to 7. There was a washout of at least 60 minutes between tasting each vehicle.
- Treatment Sequence: ABDGHEF: Sisunatovir 400 mg, Fed (treatment A) was administered Q12h for 4 days in Period 1, followed by sisunatovir 200 mg plus matching placebo, Fed (treatment B) Q12h for 4 days in Period 2 followed by sisunatovir 200 mg, Fasted (treatment D) administered Q12h for 4 days in Period 3. There was a washout period of minimum 7 days between each subsequent period. Participants tasted sisunatovir 50 mg in apple juice (treatment G) and sisunatovir 50 mg in saline (treatment H), sisunatovir 50 mg capsule content in water (treatment E), sisunatovir 50 mg in Formula (treatment F) on Day 1 of treatment period 4 to 7. There was a washout of at least 60 minutes between tasting each vehicle.
- Treatment Sequence: ACDEFGH: Sisunatovir 400 mg, Fed (treatment A) was administered Q12h for 4 days in Period 1, followed by Placebo, Fed (treatment C) Q12h for 4 days in Period 2 followed by sisunatovir 200 mg, Fasted (treatment D) administered Q12h for 4 days in Period 3. There was a washout period of minimum 7 days between each subsequent period. Participants tasted Sisunatovir 50 mg, Water (Treatment E) sisunatovir 50 mg in Formula (treatment F), sisunatovir 50 mg in apple juice (treatment G) and sisunatovir 50 mg in saline (treatment H), on Day 1 of treatment period 4 to 7. There was a washout of at least 60 minutes between tasting each vehicle.
- Treatment Sequence: ACDFGHE: Sisunatovir 400 mg, Fed (treatment A) was administered Q12h for 4 days in Period 1, followed by Placebo, Fed (treatment C) Q12h for 4 days in Period 2 followed by sisunatovir 200 mg, Fasted (treatment D) administered Q12h for 4 days in Period 3. There was a washout period of minimum 7 days between each subsequent period. Participants tasted sisunatovir 50 mg in Formula (treatment F), sisunatovir 50 mg in apple juice (treatment G), sisunatovir 50 mg in saline (treatment H), Sisunatovir 50 mg, Water (Treatment E), and on Day 1 of treatment period 4 to 7. There was a washout of at least 60 minutes between tasting each vehicle.
- Treatment Sequence: ACDGHEF: Sisunatovir 400 mg, Fed (treatment A) was administered Q12h for 4 days in Period 1, followed by Placebo, Fed (treatment C) Q12h for 4 days in Period 2 followed by sisunatovir 200 mg, Fasted (treatment D) administered Q12h for 4 days in Period 3. There was a washout period of minimum 7 days between each subsequent period. Participants tasted sisunatovir 50 mg in apple juice (treatment G), sisunatovir 50 mg in saline (treatment H), Sisunatovir 50 mg, Water (Treatment E), and sisunatovir 50 mg in Formula (treatment F) on Day 1 of treatment period 4 to 7. There was a washout of at least 60 minutes between tasting each vehicle.
- Treatment Sequence: BLDEFGH: Sisunatovir 200 mg, Fed (treatment B) was administered Q12h for 4 days in Period 1, followed by Sisunatovir 200 mg, Fed (treatment L) Q12h for 4 days in Period 2 followed by sisunatovir 200 mg, Fasted (treatment D) administered Q12h for 4 days in Period 3. There was a washout period of minimum 7 days between each subsequent period. Participants tasted sisunatovir 50 mg capsule content in water (treatment E), sisunatovir 50 mg in Formula (treatment F), sisunatovir 50 mg in apple juice (treatment G) and sisunatovir 50 mg in saline (treatment H), on Day 1 of treatment period 4 to 7. There was a washout of at least 60 minutes between tasting each vehicle.
- Treatment Sequence: BLDFGHE: Sisunatovir 200 mg, Fed (treatment B) was administered Q12h for 4 days in Period 1, followed by Sisunatovir 200 mg, Fed (treatment L) Q12h for 4 days in Period 2 followed by sisunatovir 200 mg, Fasted (treatment D) administered Q12h for 4 days in Period 3. There was a washout period of minimum 7 days between each subsequent period. Participants tasted sisunatovir 50 mg in Formula (treatment F), sisunatovir 50 mg in apple juice (treatment G) and sisunatovir 50 mg in saline (treatment H) and sisunatovir 50 mg capsule content in water (treatment E) on Day 1 of treatment period 4 to 7. There was a washout of at least 60 minutes between tasting each vehicle.
- Treatment Sequence: BLDGHEF: Sisunatovir 200 mg, Fed (treatment B) was administered Q12h for 4 days in Period 1, followed by Sisunatovir 200 mg, Fed (treatment L) Q12h for 4 days in Period 2 followed by sisunatovir 200 mg, Fasted (treatment D) administered Q12h for 4 days in Period 3. There was a washout period of minimum 7 days between each subsequent period. Participants tasted sisunatovir 50 mg in apple juice (treatment G), sisunatovir 50 mg in saline (treatment H), sisunatovir 50 mg capsule content in water (treatment E) and sisunatovir 50 mg in Formula (treatment F) on Day 1 of treatment period 4 to 7. There was a washout of at least 60 minutes between tasting each vehicle.
- Treatment Sequence: CLDEFGH: Placebo, Fed (treatment C) was administered Q12h for 4 days in Period 1, followed by Sisunatovir 200 mg, Fed (treatment L) Q12h for 4 days in Period 2 followed by sisunatovir 200 mg, Fasted (treatment D) administered Q12h for 4 days in Period 3. There was a washout period of minimum 7 days between each subsequent period. Participants tasted sisunatovir 50 mg capsule content in water (treatment E), sisunatovir 50 mg in Formula (treatment F) sisunatovir 50 mg in apple juice (treatment G) and sisunatovir 50 mg in saline (treatment H) on Day 1 of treatment period 4 to 7. There was a washout of at least 60 minutes between tasting each vehicle.
- Treatment Sequence: CLDFGHE: Placebo, Fed (treatment C) was administered Q12h for 4 days in Period 1, followed by Sisunatovir 200 mg, Fed (treatment L) Q12h for 4 days in Period 2 followed by sisunatovir 200 mg, Fasted (treatment D) administered Q12h for 4 days in Period 3. There was a washout period of minimum 7 days between each subsequent period. Participants tasted sisunatovir 50 mg in Formula (treatment F) sisunatovir 50 mg in apple juice (treatment G) and sisunatovir 50 mg in saline (treatment H) and sisunatovir 50 mg capsule content in water (treatment E) on Day 1 of treatment period 4 to 7. There was a washout of at least 60 minutes between tasting each vehicle.
- Treatment Sequence: CLDGHEF: Placebo, Fed (treatment C) was administered Q12h for 4 days in Period 1, followed by Sisunatovir 200 mg, Fed (treatment L) Q12h for 4 days in Period 2 followed by sisunatovir 200 mg, Fasted (treatment D) administered Q12h for 4 days in Period 3. There was a washout period of minimum 7 days between each subsequent period. Participants tasted sisunatovir 50 mg in apple juice (treatment G) and sisunatovir 50 mg in saline (treatment H) and sisunatovir 50 mg capsule content in water (treatment E) and sisunatovir 50 mg in Formula (treatment F) on Day 1 of treatment period 4 to 7. There was a washout of at least 60 minutes between tasting each vehicle.
Period: Part 1 Period 1 (4 Days)
Arm/Group | Treatment Sequence: ABDEFGH | Treatment Sequence: ABDFGHE | Treatment Sequence: ABDGHEF | Treatment Sequence: ACDEFGH | Treatment Sequence: ACDFGHE | Treatment Sequence: ACDGHEF | Treatment Sequence: BLDEFGH | Treatment Sequence: BLDFGHE | Treatment Sequence: BLDGHEF | Treatment Sequence: CLDEFGH | Treatment Sequence: CLDFGHE | Treatment Sequence: CLDGHEF
Started | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1 Period 2 (4 Days)
Arm/Group | Treatment Sequence: ABDEFGH | Treatment Sequence: ABDFGHE | Treatment Sequence: ABDGHEF | Treatment Sequence: ACDEFGH | Treatment Sequence: ACDFGHE | Treatment Sequence: ACDGHEF | Treatment Sequence: BLDEFGH | Treatment Sequence: BLDFGHE | Treatment Sequence: BLDGHEF | Treatment Sequence: CLDEFGH | Treatment Sequence: CLDFGHE | Treatment Sequence: CLDGHEF
Started | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1 Period 3 (4 Days)
Arm/Group | Treatment Sequence: ABDEFGH | Treatment Sequence: ABDFGHE | Treatment Sequence: ABDGHEF | Treatment Sequence: ACDEFGH | Treatment Sequence: ACDFGHE | Treatment Sequence: ACDGHEF | Treatment Sequence: BLDEFGH | Treatment Sequence: BLDFGHE | Treatment Sequence: BLDGHEF | Treatment Sequence: CLDEFGH | Treatment Sequence: CLDFGHE | Treatment Sequence: CLDGHEF
Started | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Refused further treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Part 2 Period 4 (1 Day)
Arm/Group | Treatment Sequence: ABDEFGH | Treatment Sequence: ABDFGHE | Treatment Sequence: ABDGHEF | Treatment Sequence: ACDEFGH | Treatment Sequence: ACDFGHE | Treatment Sequence: ACDGHEF | Treatment Sequence: BLDEFGH | Treatment Sequence: BLDFGHE | Treatment Sequence: BLDGHEF | Treatment Sequence: CLDEFGH | Treatment Sequence: CLDFGHE | Treatment Sequence: CLDGHEF
Started | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2 Period 5 (1 Day)
Arm/Group | Treatment Sequence: ABDEFGH | Treatment Sequence: ABDFGHE | Treatment Sequence: ABDGHEF | Treatment Sequence: ACDEFGH | Treatment Sequence: ACDFGHE | Treatment Sequence: ACDGHEF | Treatment Sequence: BLDEFGH | Treatment Sequence: BLDFGHE | Treatment Sequence: BLDGHEF | Treatment Sequence: CLDEFGH | Treatment Sequence: CLDFGHE | Treatment Sequence: CLDGHEF
Started | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2 Period 6 (1 Day)
Arm/Group | Treatment Sequence: ABDEFGH | Treatment Sequence: ABDFGHE | Treatment Sequence: ABDGHEF | Treatment Sequence: ACDEFGH | Treatment Sequence: ACDFGHE | Treatment Sequence: ACDGHEF | Treatment Sequence: BLDEFGH | Treatment Sequence: BLDFGHE | Treatment Sequence: BLDGHEF | Treatment Sequence: CLDEFGH | Treatment Sequence: CLDFGHE | Treatment Sequence: CLDGHEF
Started | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2 Period 7 (1 Day)
Arm/Group | Treatment Sequence: ABDEFGH | Treatment Sequence: ABDFGHE | Treatment Sequence: ABDGHEF | Treatment Sequence: ACDEFGH | Treatment Sequence: ACDFGHE | Treatment Sequence: ACDGHEF | Treatment Sequence: BLDEFGH | Treatment Sequence: BLDFGHE | Treatment Sequence: BLDGHEF | Treatment Sequence: CLDEFGH | Treatment Sequence: CLDFGHE | Treatment Sequence: CLDGHEF
Started | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Groups:
- All Participants: Participants who were randomized to either of the treatment sequence and received Sisunatovir 400 mg, Fed (A) Sisunatovir 200 mg, Fed (B), Placebo, Fed (treatment C), Sisunatovir 200 mg, Fasted (D), Sisunatovir 200 mg, Fed (treatment L), Sisunatovir 50 mg, Water (E), Sisunatovir 50 mg, Formula (F), Sisunatovir 50 mg, Apple Juice (G), Sisunatovir 50 mg, Saline (H) in any of the treatment periods were included. Participants were administered either Sisunatovir 200 mg in the fed state, Sisunatovir 400 mg in the fed state or placebo in fed state in Period 1 and 2, Sisunatovir 200 mg in fasted state in Period 3 and tasted Sisunatovir 50 mg capsule in either water, formula, apple juice or saline in Periods 4 to 7.
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.3 (10.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs were any AEs that occurred following start of treatment.
Time Frame: From start of treatment to 28-35 days after last dose (maximum upto 66 days)
Population: Safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants were analyzed according to the product they actually received.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Sisunatovir 400 mg, Fed: Participants were administered sisunatovir 400 mg once every 12 hours for 4 days plus 1 dose as 50 mg capsules in a fed state in either period 1 or 2 of Part 1.
- Part 1: Sisunatovir 200 mg, Fed: Participants were administered sisunatovir 200 mg once every 12 hours for 4 days plus 1 dose as 50 mg capsules in a fed state in either period 1 or 2 of Part 1.
- Part 1: Placebo, Fed: Participants were administered placebo once every 12 hours for 4 days plus 1 dose in a fed state in either period 1 or 2 of Part 1.
- Part 1: Sisunatovir 200 mg, Fasted: Participants were administered sisunatovir 200 mg once every 12 hours for 4 days plus 1 dose in a fasted state in period 3 of Part 1.
- Part 2: Sisunatovir 50 mg, Water: Participants tasted sisunatovir 50 mg capsule content in water and then spat out the drug to assess the palatability.
- Part 2: Sisunatovir 50 mg, Formula: Participants tasted sisunatovir 50 mg capsule content in formula and then spat out the drug to assess the palatability.
- Part 2: Sisunatovir 50 mg, Apple Juice: Participants tasted sisunatovir 50 mg capsule content in Apple Juice and then spat out the drug to assess the palatability.
- Part 2: Sisunatovir 50 mg, Saline: Participants tasted sisunatovir 50 mg capsule content in saline and then spat out the drug to assess the palatability.
Arm/Group | Part 1: Sisunatovir 400 mg, Fed | Part 1: Sisunatovir 200 mg, Fed | Part 1: Placebo, Fed | Part 1: Sisunatovir 200 mg, Fasted | Part 2: Sisunatovir 50 mg, Water | Part 2: Sisunatovir 50 mg, Formula | Part 2: Sisunatovir 50 mg, Apple Juice | Part 2: Sisunatovir 50 mg, Saline
Number analyzed (Participants) | 6 | 12 | 6 | 11 | 11 | 11 | 11 | 11
Participants | 6 | 7 | 4 | 9 | 2 | 1 | 0 | 2

2. Primary Outcome: Number of Participants With Clinical Laboratory Abnormalities: Part 1
Description: Laboratory tests included haematology (Monocytes [10^9/L] increase: > 1.2* upper limit of normal [ULN] and Monocytes/Leukocytes [percentage] {%}:> 1.2* ULN); clinical chemistry (serum) included Alanine Aminotransferase (units per liter [U/L]):> 3.0* ULN and Bicarbonate (milliequivalents per liter) (mEq/L): >1.1* ULN and in urinalysis (urine Hemoglobin (Scalar) more than equal to (>=) 1, urine Bilirubin (Scalar) >= 1, Hyaline Casts (/Low power field [LPF]) >= 1. Number of participants with any clinical laboratory abnormalities is reported in this outcome.
Time Frame: Up to Day 5
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Sisunatovir 400 mg, Fed: Participants were administered sisunatovir 400 mg once every 12 hours for 4 days plus 1 dose as 50 mg capsules in a fed state in either period 1 or 2 of Part 1.
- Sisunatovir 200 mg, Fed: Participants were administered sisunatovir 200 mg once every 12 hours for 4 days plus 1 dose as 50 mg capsules in a fed state in either period 1 or 2 of Part 1.
- Placebo, Fed: Participants were administered placebo once every 12 hours for 4 days plus 1 dose in a fed state in either period 1 or 2 of Part 1.
- Sisunatovir 200 mg, Fasted: Participants were administered sisunatovir 200 mg once every 12 hours for 4 days plus 1 dose in a fasted state in period 3 of Part 1.
Arm/Group | Sisunatovir 400 mg, Fed | Sisunatovir 200 mg, Fed | Placebo, Fed | Sisunatovir 200 mg, Fasted
Number analyzed (Participants) | 6 | 12 | 6 | 11
Participants | 2 | 2 | 4 | 5

3. Primary Outcome: Number of Participants With Newly Occurring Notable Abnormal Vital Signs: Part 1
Description: Supine blood pressure (BP) was measured with the participant's arm supported at the level of the heart and recorded after approximately 5 minutes of rest. Pulse rate was measured in the brachial/radial artery. Notable abnormal vital sign categories included: Systolic BP: <90 millimeter of mercury [mmHg]; Systolic BP change from baseline: maximum increase and decrease >=30 mmHg; Diastolic BP <50 mmHg; Diastolic BP change from baseline: maximum decrease and increase ≥20 mmHg; pulse rate <40 and >120 beats per minute. Number of participants with newly occurring notable abnormal vital sign (i.e. change in supine systolic BP >=30 millimeter of mercury [mmHg] increase) is reported in this outcome measure.
Time Frame: Up to Day 5
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sisunatovir 400 mg, Fed | Sisunatovir 200 mg, Fed | Placebo, Fed | Sisunatovir 200 mg, Fasted
Number analyzed (Participants) | 6 | 12 | 6 | 11
Participants | 0 | 1 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG) Findings: Part 1
Description: Standard 12-lead ECGs utilizing limb leads were used to measure PR interval, QT interval, QTc corrected using Fridericia's formula (QTcF), and QRS complex. ECG was performed after the participant had rested quietly for at least 5 minutes in a supine position. Clinical significance was determined by the investigator.
Time Frame: Up to Day 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sisunatovir 400 mg, Fed | Sisunatovir 200 mg, Fed | Placebo, Fed | Sisunatovir 200 mg, Fasted
Number analyzed (Participants) | 6 | 12 | 6 | 11
Participants | 0 | 0 | 0 | 1

5. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) for Day 1: Part 1
Description: Area under the concentration-time profile from time zero to time tau (the dosing interval), where tau = 12 hours for twice a day (BID) dosing.
Time Frame: Pre-dose, 1, 2, 3, 4, 5, 6, 8 and 12 hours post-dose on Day 1
Population: Pharmacokinetic (PK) parameter analysis population included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention and in whom at least 1 of the PK parameters of interest could be reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour/ milliliter (ng*hr/mL)
Arm/Group | Sisunatovir 400 mg, Fed | Sisunatovir 200 mg, Fed | Sisunatovir 200 mg, Fasted
Number analyzed (Participants) | 6 | 12 | 11
Nanogram*hour/ milliliter (ng*hr/mL) | 2623 (30) | 495.7 (48) | 338.4 (72)

6. Secondary Outcome: Dose Normalized AUCtau (AUCtau [dn]) for Day 1: Part 1
Description: AUCtau(dn) was calculated as AUCtau/Dose.
Time Frame: Pre-dose, 1, 2, 3, 4, 5, 6, 8 and 12 hours post-dose on Day 1
Population: PK parameter analysis population included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention and in whom at least 1 of the PK parameters of interest could be reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour/ milliliter/milligram
Arm/Group | Sisunatovir 400 mg, Fed | Sisunatovir 200 mg, Fed | Sisunatovir 200 mg, Fasted
Number analyzed (Participants) | 6 | 12 | 11
Nanogram*hour/ milliliter/milligram | 6.554 (30) | 2.478 (48) | 1.691 (72)

7. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Day 1: Part 1
Time Frame: Pre-dose, 1, 2, 3, 4, 5, 6, 8 and 12 hours post-dose on Day 1
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter (ng/mL)
Arm/Group | Sisunatovir 400 mg, Fed | Sisunatovir 200 mg, Fed | Sisunatovir 200 mg, Fasted
Number analyzed (Participants) | 6 | 12 | 11
Nanogram/milliliter (ng/mL) | 410.8 (20) | 72.00 (47) | 50.09 (77)

8. Secondary Outcome: Dose Normalized Maximum Plasma Concentration (Cmax [dn]) for Day 1: Part 1
Description: Cmax(dn) was calculated as Cmax/Dose.
Time Frame: Pre-dose, 1, 2, 3, 4, 5, 6, 8 and 12 hours post-dose on Day 1
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter/milligram (ng/mL/mg)
Arm/Group | Sisunatovir 400 mg, Fed | Sisunatovir 200 mg, Fed | Sisunatovir 200 mg, Fasted
Number analyzed (Participants) | 6 | 12 | 11
Nanogram/milliliter/milligram (ng/mL/mg) | 1.028 (20) | 0.3602 (47) | 0.2507 (77)

9. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) for Day 1: Part 1
Time Frame: Pre-dose, 1, 2, 3, 4, 5, 6, 8 and 12 hours post-dose on Day 1
Population: as for outcome 6
Measure: Median (Full Range); unit: Hour
Arm/Group | Sisunatovir 400 mg, Fed | Sisunatovir 200 mg, Fed | Sisunatovir 200 mg, Fasted
Number analyzed (Participants) | 6 | 12 | 11
Hour | 5.00 [3.00 to 5.00] | 5.00 [3.00 to 5.03] | 5.00 [4.00 to 6.00]

10. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) for Day 5: Part 1
Description: Area under the concentration-time profile from time zero to time tau (the dosing interval), where tau = 12 hours for BID dosing.
Time Frame: Pre-dose, 1, 2, 3, 4, 5, 6, 8 and 12 hours post-dose on Day 5
Population: PK parameter analysis population included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention and in whom at least 1 of the PK parameters of interest could be reported. Here, Number of Participants Analyzed' signifies participants evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour/ milliliter (ng*hr/mL)
Arm/Group | Sisunatovir 400 mg, Fed | Sisunatovir 200 mg, Fed | Sisunatovir 200 mg, Fasted
Number analyzed (Participants) | 5 | 12 | 11
Nanogram*hour/ milliliter (ng*hr/mL) | 7244 (47) | 787.6 (57) | 678.2 (51)

11. Secondary Outcome: AUCtau(dn) for Day 5: Part 1
Description: AUCtau(dn) was calculated as AUCtau/Dose.
Time Frame: Pre-dose, 1, 2, 3,4, 5, 6, 8 and 12 hours post-dose on Day 5
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour/milliliter/milligram
Arm/Group | Sisunatovir 400 mg, Fed | Sisunatovir 200 mg, Fed | Sisunatovir 200 mg, Fasted
Number analyzed (Participants) | 5 | 12 | 11
Nanogram*hour/milliliter/milligram | 18.10 (47) | 3.939 (57) | 3.388 (51)

12. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Day 5: Part 1
Time Frame: Pre-dose, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36 and 48 hours post-dose on Day 5
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter (ng/mL)
Arm/Group | Sisunatovir 400 mg, Fed | Sisunatovir 200 mg, Fed | Sisunatovir 200 mg, Fasted
Number analyzed (Participants) | 5 | 12 | 11
Nanogram/milliliter (ng/mL) | 811.0 (41) | 97.89 (52) | 76.92 (53)

13. Secondary Outcome: Cmax(dn) for Day 5: Part 1
Description: Cmax(dn) was calculated as Cmax/Dose.
Time Frame: Pre-dose, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36 and 48 hours post-dose on Day 5
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | Sisunatovir 400 mg, Fed | Sisunatovir 200 mg, Fed | Sisunatovir 200 mg, Fasted
Number analyzed (Participants) | 5 | 12 | 11
ng/mL/mg | 2.031 (41) | 0.4900 (52) | 0.3847 (53)

14. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) for Day 5: Part 1
Time Frame: Pre-dose, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36 and 48 hours post-dose on Day 5
Population: as for outcome 10
Measure: Median (Full Range); unit: Hour
Arm/Group | Sisunatovir 400 mg, Fed | Sisunatovir 200 mg, Fed | Sisunatovir 200 mg, Fasted
Number analyzed (Participants) | 5 | 12 | 11
Hour | 4.00 [3.00 to 5.00] | 5.00 [3.00 to 5.03] | 5.00 [3.00 to 6.00]

15. Secondary Outcome: Apparent Clearance (CL/F) for Day 5: Part 1
Description: CL/F was calculated as Dose/AUCtau.
Time Frame: Pre-dose, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36 and 48 hours post-dose on Day 5
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour
Arm/Group | Sisunatovir 400 mg, Fed | Sisunatovir 200 mg, Fed | Sisunatovir 200 mg, Fasted
Number analyzed (Participants) | 5 | 12 | 11
Liter/hour | 55.20 (47) | 253.9 (57) | 295.2 (50)

16. Secondary Outcome: Observed Accumulation Ratio (Rac) for AUC for Day 5: Part 1
Description: Rac for AUC was calculated as AUCtau Day5/AUCtau Day1.
Time Frame: Pre-dose, 1, 2, 3, 4, 5, 6, 8 and 12 hours post-dose on Day 1 and Pre-dose, 1, 2, 3, 4, 5, 6, 8, 12 hours post-dose on Day 5
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Sisunatovir 400 mg, Fed | Sisunatovir 200 mg, Fed | Sisunatovir 200 mg, Fasted
Number analyzed (Participants) | 5 | 12 | 11
Ratio | 2.757 (24) | 1.589 (22) | 2.003 (63)

17. Secondary Outcome: Observed Accumulation Ratio for Maximum Observed Plasma Concentration (Rac,Cmax) for Day 5: Part 1
Description: Rac,Cmax was calculated as Cmax Day5/Cmax Day1.
Time Frame: Pre-dose, 1, 2, 3, 4, 5, 6, 8 and 12 hours post-dose on Day 1 and Pre-dose, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36 and 48 hours post-dose on Day 5
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Sisunatovir 400 mg, Fed | Sisunatovir 200 mg, Fed | Sisunatovir 200 mg, Fasted
Number analyzed (Participants) | 5 | 12 | 11
Ratio | 1.961 (25) | 1.360 (25) | 1.534 (69)

18. Secondary Outcome: Plasma Decay Half-Life (t1/2) for Day 5: Part 1
Time Frame: Pre-dose, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36 and 48 hours post-dose on Day 5
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Sisunatovir 400 mg, Fed | Sisunatovir 200 mg, Fed | Sisunatovir 200 mg, Fasted
Number analyzed (Participants) | 5 | 12 | 11
Hour | 9.326 (1.2781) | 10.87 (0.96844) | 11.15 (2.0984)

19. Secondary Outcome: Apparent Volume of Distribution (Vz/F) for Day 5: Part 1
Description: Vz/F was calculated as Dose/(AUCtau * kel [Terminal phase rate constant]).
Time Frame: Pre-dose, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36 and 48 hours post-dose on Day 5
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Sisunatovir 400 mg, Fed | Sisunatovir 200 mg, Fed | Sisunatovir 200 mg, Fasted
Number analyzed (Participants) | 5 | 12 | 11
Liter | 736.1 (63) | 3962 (63) | 4676 (60)

20. Secondary Outcome: AUCtau for Day 5: Evaluation of Food Effect (Sisunatovir 200 mg Fed Versus Fasted): Part 1
Time Frame: Pre-dose, 1, 2, 3, 4, 5, 6, 8, 12 hours post-dose on Day 5
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Sisunatovir 200 mg, Fed | Sisunatovir 200 mg, Fasted
Number analyzed (Participants) | 12 | 11
ng*hr/mL | 787.6 (57) | 678.2 (51)
Statistical Analysis 1: Comparison: Sisunatovir 200 mg, Fed vs Sisunatovir 200 mg, Fasted; Test type: Other; Ratio = 126.65, 90% CI 2-sided [106.87 to 150.10] — Analysis was performed using mixed effect model with sequence, and treatment as fixed effects and participant within sequence as a random effect

21. Secondary Outcome: Cmax for Day 5: Evaluation of Food Effect (Sisunatovir 200 mg Fed Versus Fasted): Part 1
Time Frame: Pre-dose, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36 and 48 hours post-dose on Day 5
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Sisunatovir 200 mg, Fed | Sisunatovir 200 mg, Fasted
Number analyzed (Participants) | 12 | 11
ng/mL | 97.89 (52) | 76.92 (53)
Statistical Analysis 1: Comparison: Sisunatovir 200 mg, Fed vs Sisunatovir 200 mg, Fasted; Test type: Other; Ratio = 142.94, 90% CI 2-sided [117.20 to 174.32] — [estimate comment as in outcome 20, analysis 1]

22. Secondary Outcome: Assessment of Overall Liking Based on Palatability Assessment Questionnaire: Part 2
Description: Participants were required to answer the palatability attribute of overall liking by providing a mark on the colour bar. The data was rescaled to a score ranging from 0 (good) to 100 (bad), where higher scores indicated less overall liking.
Time Frame: 1 minute (immediately following dose), 5,10 and 20 minutes after tasting dose in each vehicle
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: Units on a scale
Groups:
- Sisunatovir 50 mg, Water: Participants tasted sisunatovir 50 mg capsule content in water and then spat out the drug to assess the palatability.
- Sisunatovir 50 mg, Formula: Participants tasted sisunatovir 50 mg capsule content in formula and then spat out the drug to assess the palatability.
- Sisunatovir 50 mg, Apple Juice: Participants tasted sisunatovir 50 mg capsule content in Apple Juice and then spat out the drug to assess the palatability.
- Sisunatovir 50 mg, Saline: Participants tasted sisunatovir 50 mg capsule content in saline and then spat out the drug to assess the palatability.
Arm/Group | Sisunatovir 50 mg, Water | Sisunatovir 50 mg, Formula | Sisunatovir 50 mg, Apple Juice | Sisunatovir 50 mg, Saline
Number analyzed (Participants) | 11 | 11 | 11 | 11
Units on a scale
  1 minute | 74.7 [59.38 to 90.07] | 67.9 [57.67 to 78.15] | 77.6 [66.74 to 88.53] | 65.7 [55.32 to 76.14]
  5 minutes | 78.4 [70.22 to 86.51] | 73.4 [65.44 to 81.29] | 71.9 [60.13 to 83.69] | 62.3 [51.89 to 72.66]
  10 minutes | 77.6 [70.72 to 84.55] | 73.6 [65.14 to 82.13] | 70.1 [58.76 to 81.42] | 63.0 [52.94 to 73.06]
  20 minutes | 75.0 [64.66 to 85.34] | 64.9 [57.84 to 71.98] | 69.8 [58.12 to 81.52] | 55.0 [47.82 to 62.18]

23. Secondary Outcome: Assessment of Mouth Feel Based on Palatability Assessment Questionnaire: Part 2
Description: Participants were required to answer the palatability attribute of mouth feel by providing a mark on the colour bar. The data was rescaled to a score ranging from 0 (good) to 100 (bad), where higher scores indicated worse mouth feel.
Time Frame: 1 minute (immediately following dose), 5,10 and 20 minutes after tasting dose in each vehicle
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | Sisunatovir 50 mg, Water | Sisunatovir 50 mg, Formula | Sisunatovir 50 mg, Apple Juice | Sisunatovir 50 mg, Saline
Number analyzed (Participants) | 11 | 11 | 11 | 11
Units on a scale
  1 minute | 80.9 [72.49 to 89.33] | 68.4 [59.10 to 77.62] | 66.1 [56.71 to 75.47] | 68.7 [55.14 to 82.31]
  5 minutes | 78.5 [69.91 to 87.00] | 75.4 [67.95 to 82.78] | 69.5 [61.70 to 77.39] | 70.1 [58.48 to 81.70]
  10 minutes | 76.9 [69.98 to 83.84] | 76.7 [68.65 to 84.80] | 69.8 [60.61 to 79.03] | 60.3 [49.75 to 70.80]
  20 minutes | 79.1 [71.72 to 86.46] | 69.0 [61.56 to 76.44] | 67.5 [57.89 to 77.20] | 54.5 [46.33 to 62.58]

24. Secondary Outcome: Assessment of Bitterness Based on Palatability Assessment Questionnaire: Part 2
Description: Participants were required to answer the palatability attribute of bitterness by providing a mark on the colour bar. The data was rescaled to a score ranging from 0 (good) to 100 (bad), where higher scores indicated more bitterness.
Time Frame: 1 minute (immediately following dose), 5,10 and 20 minutes after tasting dose in each vehicle
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | Sisunatovir 50 mg, Water | Sisunatovir 50 mg, Formula | Sisunatovir 50 mg, Apple Juice | Sisunatovir 50 mg, Saline
Number analyzed (Participants) | 11 | 11 | 11 | 11
Units on a scale
  1 minute | 75.3 [61.82 to 88.72] | 73.5 [63.78 to 83.13] | 76.0 [65.36 to 86.64] | 64.2 [50.88 to 77.48]
  5 minutes | 78.8 [68.51 to 89.12] | 75.0 [66.51 to 83.49] | 76.0 [67.89 to 84.11] | 59.8 [47.62 to 72.02]
  10 minutes | 76.8 [68.93 to 84.70] | 77.5 [68.71 to 86.38] | 75.9 [66.97 to 84.85] | 58.1 [46.35 to 69.84]
  20 minutes | 77.9 [70.25 to 85.57] | 68.7 [59.53 to 77.93] | 73.1 [63.37 to 82.82] | 53.5 [42.66 to 64.43]

25. Secondary Outcome: Assessment of Tongue/Mouth Burn Based on Palatability Assessment Questionnaire: Part 2
Description: Participants were required to answer the palatability attribute of tongue/mouth burn by providing a mark on the colour bar. The data was rescaled to a score ranging from 0 (good) to 100 (bad), where higher scores indicated more tongue/mouth burn.
Time Frame: 1 minute (immediately following dose), 5,10 and 20 minutes after tasting dose in each vehicle
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | Sisunatovir 50 mg, Water | Sisunatovir 50 mg, Formula | Sisunatovir 50 mg, Apple Juice | Sisunatovir 50 mg, Saline
Number analyzed (Participants) | 11 | 11 | 11 | 11
Units on a scale
  1 minute | 22.6 [5.95 to 39.32] | 17.9 [3.34 to 32.48] | 20.5 [4.84 to 36.07] | 26.3 [8.91 to 43.63]
  5 minutes | 32.6 [15.17 to 50.10] | 24.1 [6.80 to 41.38] | 21.2 [4.91 to 37.45] | 26.5 [10.37 to 42.72]
  10 minutes | 38.6 [19.62 to 57.65] | 25.0 [6.38 to 43.62] | 25.3 [5.18 to 45.37] | 24.6 [10.32 to 38.95]
  20 minutes | 35.8 [16.58 to 55.05] | 23.6 [6.64 to 40.63] | 23.1 [6.37 to 39.81] | 24.4 [10.13 to 38.60]

26. Secondary Outcome: Assessment of Sourness Based on Palatability Assessment Questionnaire: Part 2
Description: Participants were required to answer the palatability attribute of sourness by providing a mark on the colour bar. The data was rescaled to a score ranging from 0 (good) to 100 (bad), where higher scores indicated increase in sourness.
Time Frame: 1 minute (immediately following dose), 5,10 and 20 minutes after tasting dose in each vehicle
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | Sisunatovir 50 mg, Water | Sisunatovir 50 mg, Formula | Sisunatovir 50 mg, Apple Juice | Sisunatovir 50 mg, Saline
Number analyzed (Participants) | 11 | 11 | 11 | 11
Units on a scale
  1 minute | 53.5 [34.11 to 72.79] | 32.8 [13.90 to 51.74] | 45.5 [28.51 to 62.58] | 34.6 [18.47 to 50.80]
  5 minutes | 52.3 [33.83 to 70.71] | 45.5 [25.77 to 65.14] | 46.9 [28.33 to 65.49] | 28.8 [13.33 to 44.31]
  10 minutes | 49.5 [31.01 to 67.90] | 38.3 [18.12 to 58.43] | 44.0 [24.71 to 63.29] | 29.2 [13.58 to 44.79]
  20 minutes | 50.3 [34.50 to 66.05] | 35.7 [17.11 to 54.34] | 44.9 [26.06 to 63.76] | 29.1 [14.13 to 44.05]

27. Secondary Outcome: Assessment of Saltiness Based on Palatability Assessment Questionnaire: Part 2
Description: Participants were required to answer the palatability attribute of saltiness by providing a mark on the colour bar. The data was rescaled to a score ranging from 0 (good) to 100 (bad), where higher scores indicated more saltiness.
Time Frame: 1 minute (immediately following dose), 5,10 and 20 minutes after tasting dose in each vehicle
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | Sisunatovir 50 mg, Water | Sisunatovir 50 mg, Formula | Sisunatovir 50 mg, Apple Juice | Sisunatovir 50 mg, Saline
Number analyzed (Participants) | 11 | 11 | 11 | 11
Units on a scale
  1 minute | 34.8 [17.12 to 52.51] | 26.7 [10.63 to 42.83] | 36.0 [18.18 to 53.82] | 56.4 [37.57 to 75.16]
  5 minutes | 39.1 [19.22 to 58.96] | 34.8 [17.94 to 51.69] | 38.3 [19.31 to 57.24] | 49.8 [33.79 to 65.85]
  10 minutes | 33.4 [16.22 to 50.50] | 30.0 [14.55 to 45.45] | 30.6 [15.06 to 46.21] | 46.8 [31.99 to 61.65]
  20 minutes | 32.3 [15.10 to 49.44] | 32.1 [15.55 to 48.63] | 29.2 [12.27 to 46.09] | 46.8 [32.61 to 61.03]

28. Secondary Outcome: Assessment of Sweetness on Palatability Assessment Questionnaire: Part 2
Description: Participants were required to answer the palatability attribute of sweetness by providing a mark on the colour bar. The data was rescaled to a score ranging from 0 (good) to 100 (bad), Participants were required to answer the palatability attribute of sweetness by providing a mark on the colour bar. The data was rescaled to a score ranging from 0 (good) to 100 (bad), where higher scores indicated more sweetness.
Time Frame: 1 minute (immediately following dose), 5,10 and 20 minutes after tasting dose in each vehicle
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | Sisunatovir 50 mg, Water | Sisunatovir 50 mg, Formula | Sisunatovir 50 mg, Apple Juice | Sisunatovir 50 mg, Saline
Number analyzed (Participants) | 11 | 11 | 11 | 11
Units on a scale
  1 minute | 16.5 [-0.06 to 33.15] | 43.9 [27.47 to 60.35] | 36.7 [20.79 to 52.67] | 26.3 [9.24 to 43.30]
  5 minutes | 21.7 [4.00 to 39.46] | 36.6 [16.88 to 56.39] | 26.5 [11.70 to 41.39] | 25.2 [8.15 to 42.21]
  10 minutes | 20.6 [2.87 to 38.40] | 27.6 [10.16 to 45.12] | 27.6 [11.26 to 44.02] | 25.0 [8.24 to 41.76]
  20 minutes | 22.2 [3.66 to 40.70] | 33.5 [14.66 to 52.43] | 29.3 [11.63 to 46.91] | 25.3 [7.60 to 42.95]

ADVERSE EVENTS:
Time Frame: From start of treatment to 28-35 days after last dose (maximum up to 66 days).
Arm/Group | Part 1: Sisunatovir 400 mg, Fed | Part 1: Sisunatovir 200 mg, Fed | Part 1: Placebo, Fed | Part 1: Sisunatovir 200 mg, Fasted | Part 2: Sisunatovir 50 mg, Water | Part 2: Sisunatovir 50 mg, Formula | Part 2: Sisunatovir 50 mg, Apple Juice | Part 2: Sisunatovir 50 mg, Saline
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/12 | 0/6 | 0/11 | 0/11 | 0/11 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/12 | 0/6 | 0/11 | 0/11 | 0/11 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 6/6 | 7/12 | 4/6 | 9/11 | 2/11 | 1/11 | 0/11 | 2/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Sisunatovir 400 mg, Fed (N=6) | Part 1: Sisunatovir 200 mg, Fed (N=12) | Part 1: Placebo, Fed (N=6) | Part 1: Sisunatovir 200 mg, Fasted (N=11) | Part 2: Sisunatovir 50 mg, Water (N=11) | Part 2: Sisunatovir 50 mg, Formula (N=11) | Part 2: Sisunatovir 50 mg, Apple Juice (N=11) | Part 2: Sisunatovir 50 mg, Saline (N=11)
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 1 | 1 | 4 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Abnormal faeces (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 1 | 4 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 1
Oesophageal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Feeling drunk (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 3 | 1 | 0 | 0 | 0
Bradyphrenia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nightmare (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-12-23): https://cdn.clinicaltrials.gov/large-docs/60/NCT05712460/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/60/NCT05712460/SAP_001.pdf